CLINICAL TRIAL: NCT02546089
Title: Investigating the Effects of Ultrasound Guided Autologous Blood Injection for Chronic Plantar Fasciitis Versus Ultrasound Guided Dry-needling Alone, a Randomised Controlled Trial
Brief Title: ABI v Dry Needling for Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHL - 11334
Record Dates: First submitted 2015-06-15; First posted 2015-09-10 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Active Comparator): local anaesthetic - lidocaine 1%, dry needling, autologous blood injection,
  + structured rehab programme
  Interventions: Other: Autologous Blood Injection; Other: Structured rehabilitation programme; Other: dry needling injection
- control group (Placebo Comparator): local anaesthetic - lidocaine 1%, dry needling,
  + structured rehab programme
  Interventions: Other: Structured rehabilitation programme; Other: dry needling injection

INTERVENTIONS:
Other: Autologous Blood Injection — ultrasound-guided autologous blood injection procedure
  Arms: intervention group
Other: Structured rehabilitation programme — (this intervention is given to patients in both arms of the study) - a standardised structured rehabilitation programme of home exercises that the patient is instructed on how to start, and how to progress during the study period
Other: dry needling injection — (this intervention is given to patients in both arms of the study) - ultrasound-guided dry needling injection performed under ultrasound guidance

SUMMARY:
To investigate whether a procedure of ultrasound-guided autologous blood injections (ABI), which includes a dry-needling component within the overall procedure, has any measureable clinical benefit over ultrasound-guided dry needling alone in patients with chronic plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 or over who are being seen in the Department of Sports Medicine (all of whom are age 16 or over) with chronic plantar fasciitis of at least 6 months duration
2. Failure of previous conservative therapy - including physiotherapy, and podiatry input
3. Objective evidence of plantar fasciitis - either ultrasound or MRI investigations
4. No contraindications of injection therapy - anticoagulation, blood borne illness, strong needle phobia …

Exclusion Criteria:

1. Patients with either partial or full-thickness tears of plantar fascia found on investigations
2. Subjects who are unable to give valid consent for study entry based on normal competency assessment
3. Subjects unable or unwilling to undergo the rehabilitation plan post-procedure
4. Subjects unable or unwilling to attend the follow-up appointments post-procedure

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Reduction in pain - as assessed by 0-10 VAS scale | 3 & 6 months - primary outcome set at 6 months for study, but using 3 month interim result as well

SECONDARY OUTCOMES:
Reduction in pain / improvement in function - as assessed by several PROMS (as below) | 3 & 6 months
  validated PROMs in use in this study include: FFI-r, MOXFQ, FAAM

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wheeler, Principal Investigator — UHL NHS Trust
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom